CLINICAL TRIAL: NCT06635889
Title: Double-Blind Randomized Placebo Controlled Trial of Intravesical Bupivacaine on Post-Operative Ureteroscopy Pain
Brief Title: Intravesical Bupivacaine on Post-Operative Ureteroscopy Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB24-1600
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Nephrolithiasis
MeSH Terms: conditions — Nephrolithiasis | interventions — Bupivacaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 50 ml of 0.25% bupivacaine (Experimental)
  Interventions: Drug: Bupivacaine
- placebo of 50 ml of Normal Saline (Placebo Comparator)
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Bupivacaine — The dose plan is to use 50 ml of 0.25% bupivacaine which corresponds with a total dose of 125mg.
  Arms: 50 ml of 0.25% bupivacaine
Other: Normal saline — Placebo of 50 ml of Normal Saline
  Arms: placebo of 50 ml of Normal Saline

SUMMARY:
Post-operative pain and lower urinary tract symptoms are common following ureteroscopy in the treatment of stone disease. The use of bupivacaine as a topical pain medication is used routinely for other urologic procedures, however, to date there are no studies that have rigorously investigated the effect of instilling bupivacaine in the bladder following ureteroscopy.

This is a randomized study that will investigate the effect of instilling bupivacaine in the bladder following routine ureteroscopy, laser lithotripsy and ureteral stenting in the treatment of stone disease. Compared to a placebo of Normal Saline, our study hypothesizes that administration of topical bupivacaine in the bladder will decrease post-operative pain and lower urinary tract symptoms while improving quality of life in the early post-operative period.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study.
* Male or female, aged ≥ 18 years old.
* Diagnosis of nephrolithiasis planned for flexible or semi-rigid ureteroscopy in the treatment of stone disease with ureteral stenting.

Exclusion Criteria:

* Foley catheterization
* History of allergy to bupivacaine
* Antegrade ureteroscopy
* Transplant or ectopic kidney
* Ureteral or bladder reconstruction
* Pregnancy (which is a contraindication to elective ureteroscopy)
* Dialysis
* Surgical complication (significant bleeding, ureteral perforation, significant urothelial damage)
* Suspicion of untreated urinary tract infection
* History of pelvic radiation
* Neurologic disease with a diagnosis of neurogenic bladder dysfunction
* History of chronic pain (fibromyalgia, interstitial cystitis, opioid abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain as determined by the score on a Visual Analog Scale (VAS) upon emergence from anesthesia | At 30 minutes post-emergence, 60 minutes post-emergence, 6 hours post-emergence and on post-operative day 1
  Pain will be assessed using a Likert 10-point scale upon emergence from anesthesia in the recovery room, post-emergence 30 minutes, 60 minutes post-emergence and 6 and 24 hours post-emergence. These types of scales are commonly used to measure post operative pain both in anesthesia and in endourology

SECONDARY OUTCOMES:
Milliequivalent of morphine consumed | From Baseline to post- operative day 5
Number of bladder spasms | From Baseline to post- operative day 5
Time to void | From Baseline to post- operative day 5
Time to discharge | From Baseline to post- operative day 5
Quality of life based on the Ureteral Stent Symptom Questionnaire (USSQ) | From Baseline to post- operative day 5
  A validated tool of 38 questions that assesses the symptoms and quality of life impact of ureteral stents.
The Patient-Reported Outcomes Measurement Information System (PROMIS) Adult Function Short Form | From Baseline to post- operative day 5
Adverse events | From Baseline to post- operative day 5

CONTACTS AND LOCATIONS:
Overall Officials: Luke Reynolds, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medical Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No